CLINICAL TRIAL: NCT02885571
Title: Can Objective Compliance Monitoring Increase Mandibular Advancement Device Usage in Obstructive Sleep Apnea Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to suggestions of IRB committee in our institution
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Woo Shin, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: D-1510-035-709
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAD for subjective compliance (Active Comparator): MAD for subjective compliance group wears the same SomnoDent Flex with DentiTrac to objective group, but they are subjected to be prescribed based on the subjective compliance data, which are acquired from patient's explanation. Compliance (average daily time,
  Interventions: Device: SomnoDent Flex with DentiTrac
- MAD for objective compliance (Experimental): MAD for objective compliance group wears the same SomnoDent Flex with DentiTrac to subjective group, but they are subjected to be prescribed based on the objective compliance data, which are acquired from data recorded within SomnoDent Flex with DentiTrac.
  Interventions: Device: SomnoDent Flex with DentiTrac

INTERVENTIONS:
Device: SomnoDent Flex with DentiTrac

SUMMARY:
This study evaluates whether objective compliance monitoring can increase mandibular advancement device (MAD) usage in obstructive sleep apnea (OSA) patients. Half of participants will be assigned to objective compliance monitoring group (experimental group), while the other will be assigned to subjective compliance monitoring group (control group). A physician will prescribe and explain to patients based on data from objective or subjective compliance monitoring.

DETAILED DESCRIPTION:
The design of this study is a randomized controlled trial. Total 40 participants are randomly divided into 2 groups: objective compliance monitoring (n=20) and subjective compliance monitoring (n=20). Both groups wear the same MAD (commercial name: SomnoDent Flex with DentiTrac). They visit Seol National University Hospital at 1, 3, and 6 month after the initiation of MAD. A research coordinator acquires data by downloading from the MAD or by asking the patients, and then transfer the information to the physician. If the patient belongs to objective compliance group, data from the MAD will be transferred to the physician. But if the patient belongs to subjective compliance group, data acquired by asking patients will be transferred to the physician. A physician will prescribe and explain to patients based on data from objective or subjective compliance monitoring.The primary aims is to examine the effectiveness of SomnoDent Flex with DentiTrac, in terms of compliance.

ELIGIBILITY:
Inclusion Criteria:

* obstructive sleep apnea patients without a history of soft palate surgery and moderate to severe periodontal disease.

Exclusion Criteria:

* central sleep apnea
* active mandibular disease
* tooth grinding
* moderate to severe periodontal disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Average daily use (hours) | one month
  The average number of hours the patient wore and did not wear the SomnoDent Flex with DentiTrac for previous one month

SECONDARY OUTCOMES:
Days used for ≥ 15 min | one month
  Days the patient wore for ≥ 15 min the SomnoDent Flex with DentiTrac for previous one month
Days used for ≥ 4 hrs | one month
  Days the patient wore for ≥ 4 hrs the SomnoDent Flex with DentiTrac for previous one month

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Bin Won, Dr., Study Chair — Department of Otorhinolaryngology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips CL, Grunstein RR, Darendeliler MA, Mihailidou AS, Srinivasan VK, Yee BJ, Marks GB, Cistulli PA. Health outcomes of continuous positive airway pressure versus oral appliance treatment for obstructive sleep apnea: a randomized controlled trial. Am J Respir Crit Care Med. 2013 Apr 15;187(8):879-87. doi: 10.1164/rccm.201212-2223OC. PMID 23413266
- [Background] Kushida CA, Morgenthaler TI, Littner MR, Alessi CA, Bailey D, Coleman J Jr, Friedman L, Hirshkowitz M, Kapen S, Kramer M, Lee-Chiong T, Owens J, Pancer JP; American Academy of Sleep. Practice parameters for the treatment of snoring and Obstructive Sleep Apnea with oral appliances: an update for 2005. Sleep. 2006 Feb;29(2):240-3. doi: 10.1093/sleep/29.2.240. PMID 16494092
- [Background] Vanderveken OM, Dieltjens M, Wouters K, De Backer WA, Van de Heyning PH, Braem MJ. Objective measurement of compliance during oral appliance therapy for sleep-disordered breathing. Thorax. 2013 Jan;68(1):91-6. doi: 10.1136/thoraxjnl-2012-201900. Epub 2012 Sep 19. PMID 22993169